CLINICAL TRIAL: NCT06825195
Title: Evaluation of Fingertip Precision Pinch Force During Carrying in Fibromyalgia Patients.
Brief Title: Evaluation of Fingertip Precision Pinch Force in Fibromyalgia Patients
Status: Completed | Type: Observational
Sponsor: Dilara Ekici Zincirci (Other)
Responsible Party: Sponsor-Investigator, Dilara Ekici Zincirci, Medical doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Other Study IDs: Fibromiyalgia1
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia; Force Measurement; Isokinetic; Muscle Strength
Keywords: Fibromiyalgia; Muscle Strength; Fatigue
MeSH Terms: conditions — Fibromyalgia; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fibromiyalgia: Fibromiyalgia Patients
  Interventions: Other: isokinetic muscle strength measurement; Other: Minimum pinch force measurement
- Healthy Control: Healthy control group
  Interventions: Other: isokinetic muscle strength measurement; Other: Minimum pinch force measurement

INTERVENTIONS:
Other: isokinetic muscle strength measurement — Wrist isokinetic eccentric flexor and extensor peak Torque and fatigue will be measured at the angular velocity of 180°/s
Other: Minimum pinch force measurement — the minimum fingertip pinch force required to hold a constant weight will be measured

SUMMARY:
This study aims to evaluate the force used by fibromyalgia patients during a task compared to healthy volunteers and to evaluate its relationship with fatigue seen in these patients.

DETAILED DESCRIPTION:
Fatigue is a common symptom in fibromyalgia patients and it is known that these patients have decreased muscle strength compared to healthy volunteers. The aim of this study was to evaluate whether the minimum force to be applied during carrying is different in fibromyalgia patients compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

-Female patients diagnosed with fibromyalgia between the ages of 18-70

Exclusion Criteria:

* Those whose treatment has been changed in the last month
* Those with shoulder, elbow, wrist and hand diseases that may cause pain in the dominant upper extremity
* Those with carpal or cubital tunnel syndrome
* Those with a history of orthopedic surgery in the dominant extremity
* Those with uncontrolled metabolic disease
* Those with B12 deficiency

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Female patients with fibromyalgia diagnosis and no accompanying rheumatological disease
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
minimum pinch force | November 2024- January 2025
  minimum fingertip pinch force required to hold a constant weight
maximum pinch force | November 2024- January 2025
  maximum fingertip pinch force required to hold a constant weight
% Minimum/maksimum pinch force | November 2024- January 2025
  percentage of minimum holding force to maximum holding force

SECONDARY OUTCOMES:
isokinetik muscle strength | November 2024- January 2025
  Wrist isokinetic extensor and flexor peak torque at 180 degrees/sec

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu Şehir Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No